CLINICAL TRIAL: NCT05575024
Title: Real-time Monitoring of Hemodynamic Stability in Septic Shock Patients Undergoing Continuous Renal Replacement Therapy: Propensity Score-matched Comparison Between oXiris and Polysulfone Membranes
Brief Title: Hemodynamic Stability in Septic Shock Patients Undergoing Continuous Renal Replacement Therapy With oXiris Membrane
Acronym: HISTORIX
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Seok Han, MD, Associate Professor, Seoul National University Hospital
Other Study IDs: 2021-4067
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury Due to Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Septic AKI: Patients with septic acute kidney injury requiring continuous renal replacement therapy
  Interventions: Device: oXiris membrane; Device: Polysulfone membrane

INTERVENTIONS:
Device: oXiris membrane — Perform continuous renal replacement therapy with oXiris membrane
Device: Polysulfone membrane — Perform continuous renal replacement therapy with polysulfone membrane

SUMMARY:
The new adsorbing membrane for continuous renal replacement therapy (CRRT), oXiris, can reduce plasma cytokines and endotoxins in septic shock patients with severe acute kidney injury, compared with standard membranes. However, its hemodynamic stability or benefits have not been thoroughly evaluated although this is reasonable.

DETAILED DESCRIPTION:
The new adsorbing membrane for continuous renal replacement therapy (CRRT), oXiris, can reduce plasma cytokines and endotoxins in patients with severe acute kidney injury or sepsis, compared with standard membranes. Based on this benefit, the use of oXiris may confer better outcomes than other membranes.

The patient outcomes include cardiovascular, respiratory, renal, and overall survivals, but this information of oXiris are insufficient. Although cytokine and endotoxin removal rates are great in oXiris, the beneficial effects on the hard outcomes are needed to use oXiris in real clinical practice.

The inflammatory and cardiovascular systems have intensive crosstalk, and thus if there are remission in inflammatory process, the patients can have hemodynamic stability. Regarding this, the investigators would like to compare the hemodynamic stability between oXiris and other standard membrane such as polysulfone, using our new real-time monitoring registry.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Sepsis related acute kidney injury requiring continuous renal replacement therapy

Exclusion Criteria:

• No monitoring of blood pressure and ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have severe acute kidney injury and require continuous renal replacement therapy because of hemodynamic instability.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality | 28 days
  Risk of all-cause mortality
Occurrence rates of ventricular tachycardia, intradialytic hypotension | 28 days
  Risk of ventricular tachycardia, intradialytic hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Seung Seok Han, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No